CLINICAL TRIAL: NCT01963260
Title: A Two-Part, Single Rising Dose Study to Assess the Safety, Pharmacokinetics and Pharmacodynamics of MK-8723 in Healthy Adults and Patients With Immune Thrombocytopenia Purpura
Brief Title: Single Rising Dose Study of MK-8723 in Healthy Participants and Participants With Immune Thrombocytopenia Purpura (MK-8723-001)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8723-001
Record Dates: First submitted 2013-10-11; First posted 2013-10-16 (Estimated); Results first posted 2017-03-21 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2019-02

CONDITIONS: Immune Thrombocytopenia Purpura

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (10):
- Part 1: MK-8723 1 mg/kg in Healthy Participants (Experimental): MK-8723 1 mg/kg administered as a single IV infusion to healthy participants in Part 1.
  Interventions: Drug: MK-8723
- Part 1: MK-8723 3 mg/kg in Healthy Participants (Experimental): MK-8723 3 mg/kg administered as a single IV infusion to healthy participants in Part 1.
  Interventions: Drug: MK-8723
- Part 1: MK-8723 10 mg/kg in Healthy Participants (Experimental): MK-8723 10 mg/kg administered as a single IV infusion to healthy participants in Part 1.
  Interventions: Drug: MK-8723
- Part 1: MK-8723 30 mg/kg in Healthy Participants (Experimental): MK-8723 30 mg/kg administered as a single IV infusion to healthy participants in Part 1.
  Interventions: Drug: MK-8723
- Part 1: MK-8723 100 mg/kg in Healthy Participants (Experimental): MK-8723 100 mg/kg administered as a single IV infusion to healthy participants in Part 1.
  Interventions: Drug: MK-8723
- Part 1: Matching Placebo to MK-8723 (Placebo Comparator): Matching placebo to MK-8723 administered as a single IV infusion to healthy participants in Part 1.
  Interventions: Drug: Matching Placebo
- Part 2: MK-8723 10 mg/kg in ITP Participants (Experimental): MK-8723 10 mg/kg administered as a single IV infusion to participants with ITP in Part 2.
  Interventions: Drug: MK-8723
- Part 2: MK-8723 30 mg/kg in ITP Participants (Experimental): MK-8723 30 mg/kg administered as a single IV infusion to participants with ITP in Part 2.
  Interventions: Drug: MK-8723
- Part 2: MK-8723 100 mg/kg in ITP Participants (Placebo Comparator): MK-8723 100 mg/kg administered as a single IV infusion to participants with ITP in Part 2.
  Interventions: Drug: MK-8723
- Part 2: Matching Placebo to MK-8723 (Placebo Comparator): Matching placebo to MK-8723 administered as a single IV infusion to participants with ITP in Part 2.
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: MK-8723 — MK-8723 administered as a single IV infusion over approximately 4 hours on Day 1.
  Arms: Part 1: MK-8723 1 mg/kg in Healthy Participants; Part 1: MK-8723 10 mg/kg in Healthy Participants; Part 1: MK-8723 100 mg/kg in Healthy Participants; Part 1: MK-8723 3 mg/kg in Healthy Participants; Part 1: MK-8723 30 mg/kg in Healthy Participants; Part 2: MK-8723 10 mg/kg in ITP Participants; Part 2: MK-8723 100 mg/kg in ITP Participants; Part 2: MK-8723 30 mg/kg in ITP Participants
Drug: Matching Placebo — Matching placebo to MK-8723 administered as a single IV infusion over approximately 4 hours on Day 1.
  Arms: Part 1: Matching Placebo to MK-8723; Part 2: Matching Placebo to MK-8723

SUMMARY:
The primary objectives of this study are to assess the safety and tolerability of single rising doses of MK-8723 in healthy adult participants and adult participants with chronic immune thrombocytopenia purpura (ITP) and to assess pharmacodynamics of MK-8723 in participants with ITP. The primary hypothesis is that the true placebo-adjusted platelet response rate to MK-8723 in adult patients with chronic ITP is >50%.

DETAILED DESCRIPTION:
In Part 1 of the trial, safety and pharmacokinetics of MK-8723 will be evaluated in healthy participants. In Part 2 of the trial, safety, pharmacokinetics, and pharmacodynamics will be evaluated among participants with ITP. In Part 1, dose escalation will occur in up to 5 serial panels of participants; each participant will receive a single intravenous (IV) dose of MK-8723 (or placebo). In Part 2, dose escalation will occur in up to 3 serial panels of participants with ITP; each participant will receive a single IV dose of MK-8723 (or placebo), once safety and tolerability of the corresponding dose is shown in Part 1. Amendment 3 specified a re-enrollment procedure for eligible participants in Part 2 to participate in more than one dosing panel.

ELIGIBILITY:
Inclusion Criteria (Part 1):

* Female participants must be non-pregnant, non-breast feeding, and of non-childbearing potential
* Has a Body Mass Index (BMI) <=32 kg/m^2
* Has a body weight >= 50 kg and <= 100 kg
* Has been judged to be in good health based on medical history, physical examination, vital sign measurements, electrocardiogram (ECG), and laboratory safety tests
* Non-smoker or has not used nicotine or nicotine-containing products for at least 3 months

Inclusion Criteria (Part 2):

* Has been diagnosed with ITP at least 3 months prior
* Female ITP participants must be non-pregnant, non-breast feeding, and either of 1) non-childbearing potential or 2) must have serum beta human chorionic gonadotropin (HCG) level consistent with a non-pregnant state, and agree to use acceptable contraception from pretrial period until 84 days postdose
* Has a BMI <=36 kg/m^2
* Has been judged to be in good health, other than ITP diagnosis, based on medical history, physical examination, vital sign measurements, ECG, and laboratory safety tests

Exclusion Criteria (Part 1):

* Has a history or clinically significant endocrine, gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary, or major neurological abnormalities or diseases
* Has a history of cancer (malignancy)
* Has a history of significant multiple and/or severe allergies or has had an anaphylactic reaction or significant intolerability to prescription or non-prescription drugs or food
* Is positive for hepatitis B surface antigen, hepatitis C antibodies, or human immunodeficiency virus (HIV)
* Has had major surgery or donated or lost 1 unit of blood in the 4 weeks prior
* Has participated in another investigational trial within 4 weeks (12 weeks for biologics)
* Has received a live virus vaccination within 42 days or plans to receive such while participating in the trial
* Is unable to refrain from or anticipates the use of any medication, including prescription and non-prescription drugs and herbal remedies from 2 weeks prior and for the duration of the trial
* Consumes greater than 3 glasses of alcoholic beverages per day
* Consumes greater than 6 servings of caffeine-containing beverages per day
* Is currently a regular user of any illicit drugs or has a history of drug and/or alcohol abuse within 3 months
* Has a history of ITP or other autoimmune disease
* Has an active infection that is clinically significant

Exclusion Criteria (Part 2):

* Has a comorbid and significant hematological or immunological disorder
* Has a history of significant multiple and/or severe allergies or has had an anaphylactic reaction or significant intolerability to prescription or non-prescription drugs or food
* Is positive for hepatitis B surface antigen, hepatitis C antibodies, or HIV
* Has had major surgery or donated or lost 1 unit of blood within 4 weeks
* Has participated in another investigational trial within 4 weeks (12 weeks for biologics), excluding prior participation in the current study
* Has a history of ITP unresponsive to intravenous immunoglobulin (IVIG)
* Has had systemic corticosteroid use within 1 month (with the exception of stable low dose oral corticosteroids)
* Has had systemic IVIG or other systemic immunomodulatory therapy, excluding MK-8723 administration in the current study, within 3 months
* Has received a thrombopoietin receptor antagonist within 3 months
* Is unable to refrain from using thrombopoietin receptor agonists and/or systemic immune modulatory medications throughout the study
* Has received a live virus vaccine within 42 days prior or plans to receive such during the trial
* Consumes greater than 3 alcoholic beverages per day
* Consumes greater than 6 servings of caffeine-containing beverages per day
* Is currently a regular user of any illicit drugs or has a history of drug and/or alcohol abuse within 3 months
* Has clinical evidence of bleeding or coagulopathy including petechial rash, easy bruising, or excessive gingival bleeding with routine dental hygiene
* Has an active infection that is clinically significant

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-10-31 (Actual); Primary Completion 2015-04-26 (Actual); Study Completion 2015-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Amendment 3 specified a re-enrollment procedure for eligible participants in Part 2 to participate in more than one dosing panel.
Pre-assignment Details: 2 participants that completed Part 2 10 mg/kg were re-enrolled in Part 2 100 mg/kg & dosed. Both participants completed Part 2 100 mg/kg. 1 participant originally assigned to Part 2 30 mg/kg received placebo in error & is included in Part 2 Placebo.
Groups:
- Part 2: MK-8723 10 mg/kg in ITP Participants: MK-8723 10 mg/kg administered as a single IV infusion to participants with immune thrombocytopenia purpura (ITP) in Part 2. 2 participants were subsequently enrolled in Part 2 MK-8723 100 mg/kg.
- Part 2: MK-8723 100 mg/kg in ITP Participants: MK-8723 100 mg/kg administered as a single IV infusion to participants with ITP in Part 2. 2 participants with ITP from Part 2 MK-8723 10 mg/kg were re-enrolled into Part 2 100 mg/kg and dosed (not shown).
Period: Overall Study
Arm/Group | Part 1: MK-8723 1 mg/kg in Healthy Participants | Part 1: MK-8723 3 mg/kg in Healthy Participants | Part 1: MK-8723 10 mg/kg in Healthy Participants | Part 1: MK-8723 30 mg/kg in Healthy Participants | Part 1: MK-8723 100 mg/kg in Healthy Participants | Part 1: Matching Placebo to MK-8723 | Part 2: MK-8723 10 mg/kg in ITP Participants | Part 2: MK-8723 30 mg/kg in ITP Participants | Part 2: MK-8723 100 mg/kg in ITP Participants | Part 2: Matching Placebo to MK-8723
Started | 6 | 6 | 6 | 6 | 6 | 10 | 3 | 2 | 1 | 4
Treated | 6 | 6 | 6 | 6 | 6 | 10 | 3 | 2 | 1 | 4
Completed | 4 | 6 | 6 | 5 | 4 | 10 | 3 | 2 | 1 | 4
Not Completed | 2 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are presented for all participants that enrolled in the study according to the actual treatment administered (i.e., as treated). 2 participants that completed Part 2 MK-8723 10 mg/kg were re-enrolled in Part 2 MK-8723 100 mg/kg and dosed per protocol procedure.
Groups:
- Part 2: MK-8723 10 mg/kg in ITP Participants: MK-8723 10 mg/kg administered as a single IV infusion to participants with ITP in Part 2. 2 participants subsequently enrolled in Part 2 MK-8723 100 mg/kg.
- Part 2: MK-8723 100 mg/kg in ITP Participants: MK-8723 100 mg/kg administered as a single IV infusion to participants with ITP in Part 2. This group includes 2 participants that re-enrolled from Part 2 MK-8723 10 mg/kg.
- Total: Total of all reporting groups
Arm/Group | Part 1: MK-8723 1 mg/kg in Healthy Participants | Part 1: MK-8723 3 mg/kg in Healthy Participants | Part 1: MK-8723 10 mg/kg in Healthy Participants | Part 1: MK-8723 30 mg/kg in Healthy Participants | Part 1: MK-8723 100 mg/kg in Healthy Participants | Part 1: Matching Placebo to MK-8723 | Part 2: MK-8723 10 mg/kg in ITP Participants | Part 2: MK-8723 30 mg/kg in ITP Participants | Part 2: MK-8723 100 mg/kg in ITP Participants | Part 2: Matching Placebo to MK-8723 | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 10 | 3 | 2 | 3 | 4 | 52
Age, Continuous [Mean (Standard Deviation); unit: Years] | 25.7 (2.7) | 32.7 (13.0) | 31.0 (12.2) | 25.7 (4.2) | 32.7 (10.5) | 30.1 (9.5) | 38.7 (22.3) | 53.0 (4.2) | 38.3 (22.7) | 50.3 (13.5) | 33.2 (13.0)
Age, Customized [Number; unit: Participants]
  Between 18 and 65 years | 6 | 6 | 6 | 6 | 6 | 10 | 3 | 2 | 3 | 3 | 51
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 2 | 2 | 3 | 10
  Male | 6 | 6 | 5 | 6 | 6 | 9 | 2 | 0 | 1 | 1 | 42

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing an Adverse Event
Description: An AE is defined as any unfavorable and unintended medical occurrence in a clinical investigation participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment.
Time Frame: Up to 84 days
Population: The All Participants as Treated (APaT) population consisting of all participants who received at least one dose of study drug was used for the safety analysis.
Measure: Number; unit: Participants
Arm/Group | Part 1: MK-8723 1 mg/kg in Healthy Participants | Part 1: MK-8723 3 mg/kg in Healthy Participants | Part 1: MK-8723 10 mg/kg in Healthy Participants | Part 1: MK-8723 30 mg/kg in Healthy Participants | Part 1: MK-8723 100 mg/kg in Healthy Participants | Part 1: Matching Placebo to MK-8723 | Part 2: MK-8723 10 mg/kg in ITP Participants | Part 2: MK-8723 30 mg/kg in ITP Participants | Part 2: MK-8723 100 mg/kg in ITP Participants | Part 2: Matching Placebo to MK-8723
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 10 | 3 | 2 | 3 | 4
Participants | 2 | 2 | 4 | 1 | 4 | 6 | 1 | 2 | 2 | 2

2. Primary Outcome: Number of Participants Discontinuing Study Due to an Adverse Event (AE)
Description: as for outcome 1
Time Frame: Up to 84 Days
Population: The APaT population consisting of all participants who received at least one dose of study drug was used for the safety analysis.
Measure: Number; unit: Participants
Arm/Group | Part 1: MK-8723 1 mg/kg in Healthy Participants | Part 1: MK-8723 3 mg/kg in Healthy Participants | Part 1: MK-8723 10 mg/kg in Healthy Participants | Part 1: MK-8723 30 mg/kg in Healthy Participants | Part 1: MK-8723 100 mg/kg in Healthy Participants | Part 1: Matching Placebo to MK-8723 | Part 2: MK-8723 10 mg/kg in ITP Participants | Part 2: MK-8723 30 mg/kg in ITP Participants | Part 2: MK-8723 100 mg/kg in ITP Participants | Part 2: Matching Placebo to MK-8723
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 10 | 3 | 2 | 3 | 4
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With a Positive Platelet Response to MK-8723
Description: In participants with ITP, platelet response is a rapid, sensitive, and highly qualitative measure of response to anti-inflammatory therapy. A positive platelet response was defined as: 1) A doubling of platelet counts at the time point of maximum response (through Day 14) as compared to Day 0 AND an increase to an absolute level of ≥50,000/μL in participants with a baseline platelet count of <50,000/μL, OR 2) A 50% increase in the platelet count at the time point of maximum response (through Day 14) as compared to Day 0 in participants with a baseline platelet count of ≥50,000/μL. The analysis was specified only for participants with ITP (Part 2) that received treatment with MK-8723 or matching placebo.
Time Frame: Up to Day 14
Population: The per protocol population consisting of all participants in compliance with the protocol (e.g., availability of measurements, absence of major protocol violations) was used for the pharmacodynamic (platelet response) analysis.
Measure: Number; unit: Participants
Arm/Group | Part 2: MK-8723 10 mg/kg in ITP Participants | Part 2: MK-8723 30 mg/kg in ITP Participants | Part 2: MK-8723 100 mg/kg in ITP Participants | Part 2: Matching Placebo to MK-8723
Number analyzed (Participants) | 3 | 2 | 3 | 4
Participants | 0 | 0 | 0 | 0

4. Secondary Outcome: Area Under the Concentration-time Curve of MK-8723 From Time 0 to Infinity (AUC0-∞) Among Healthy Participants and Participants With ITP
Description: AUC0-∞ is a measure of total body exposure to drug. Serum samples for determination of AUC0-∞ were collected at pre-specified time-points.
Time Frame: All dose groups: Predose and 4 (end of infusion), 6, 12, 24 hrs postdose and Days 3, 4, 5, 7, 10, 14, 21, 28; 30 mg/kg and 100 mg/kg dose groups: Days 43, 56, 71, 84
Population: The per protocol population consisting of all participants in compliance with the protocol (e.g., availability of measurements, absence of major protocol violations) was used for the pharmacokinetic (AUC0-∞) analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*μg/mL
Arm/Group | Part 1: MK-8723 1 mg/kg in Healthy Participants | Part 1: MK-8723 3 mg/kg in Healthy Participants | Part 1: MK-8723 10 mg/kg in Healthy Participants | Part 1: MK-8723 30 mg/kg in Healthy Participants | Part 1: MK-8723 100 mg/kg in Healthy Participants | Part 2: MK-8723 10 mg/kg in ITP Participants | Part 2: MK-8723 30 mg/kg in ITP Participants | Part 2: MK-8723 100 mg/kg in ITP Participants
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 3 | 2 | 3
hr*μg/mL | 4830 (22.1) | 22300 (21.9) | 65800 (13.4) | 186000 (7.28) | 711000 (50.5) | 66200 (57.9) | 203000 (22.6) | 668000 (19.4)

5. Secondary Outcome: Maximum Concentration (Cmax) of MK-8723 Among Healthy Participants and Participants With ITP
Description: Serum samples for determination of Cmax were collected at pre-specified time-points.
Time Frame: as for outcome 4
Population: The per protocol population consisting of all participants in compliance with the protocol (e.g., availability of measurements, absence of major protocol violations) was used for this pharmacokinetic (Cmax) analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Part 1: MK-8723 1 mg/kg in Healthy Participants | Part 1: MK-8723 3 mg/kg in Healthy Participants | Part 1: MK-8723 10 mg/kg in Healthy Participants | Part 1: MK-8723 30 mg/kg in Healthy Participants | Part 1: MK-8723 100 mg/kg in Healthy Participants | Part 2: MK-8723 10 mg/kg in ITP Participants | Part 2: MK-8723 30 mg/kg in ITP Participants | Part 2: MK-8723 100 mg/kg in ITP Participants
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 3 | 2 | 3
μg/mL | 18.7 (11.4) | 72.3 (8.53) | 225 (15.5) | 844 (12.2) | 2160 (23.9) | 195 (11.7) | 741 (24.8) | 2450 (8.63)

ADVERSE EVENTS:
Time Frame: Up to 84 days
Description: The APaT population consisting of all participants who received at least one dose of study drug was used for the safety analysis. AEs are presented according to the actual treatment administered (i.e., as treated). 2 participants that completed Part 2 MK-8723 10 mg/kg were re-enrolled in Part 2 MK-8723 100 mg/kg & dosed per protocol procedure.
Arm/Group | Part 1: MK-8723 1 mg/kg in Healthy Participants | Part 1: MK-8723 3 mg/kg in Healthy Participants | Part 1: MK-8723 10 mg/kg in Healthy Participants | Part 1: MK-8723 30 mg/kg in Healthy Participants | Part 1: MK-8723 100 mg/kg in Healthy Participants | Part 1: Matching Placebo to MK-8723 | Part 2: MK-8723 10 mg/kg in ITP Participants | Part 2: MK-8723 30 mg/kg in ITP Participants | Part 2: MK-8723 100 mg/kg in ITP Participants | Part 2: Matching Placebo to MK-8723
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/10 | 0/3 | 0/2 | 0/3 | 0/4
Other Adverse Events (participants affected / at risk) | 2/6 | 2/6 | 4/6 | 1/6 | 4/6 | 6/10 | 1/3 | 2/2 | 2/3 | 2/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: MK-8723 1 mg/kg in Healthy Participants (N=6) | Part 1: MK-8723 3 mg/kg in Healthy Participants (N=6) | Part 1: MK-8723 10 mg/kg in Healthy Participants (N=6) | Part 1: MK-8723 30 mg/kg in Healthy Participants (N=6) | Part 1: MK-8723 100 mg/kg in Healthy Participants (N=6) | Part 1: Matching Placebo to MK-8723 (N=10) | Part 2: MK-8723 10 mg/kg in ITP Participants (N=3) | Part 2: MK-8723 30 mg/kg in ITP Participants (N=2) | Part 2: MK-8723 100 mg/kg in ITP Participants (N=3) | Part 2: Matching Placebo to MK-8723 (N=4)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Frequent bowel movements (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Feeling abnormal (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Infectious mononucleosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 5 (6) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia intercostal (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results.